CLINICAL TRIAL: NCT00486447
Title: A Prospective Multi-center Study Comparing Cardiac Computed Tomography (CT) Using a 64-detector Row Volumetric Computed Tomography (VCT) Scanner for the Detection of Coronary Artery Disease With Cardiac Radionuclide Imaging.
Brief Title: Perfusion Imaging and CT -Understanding Relative Efficacy
Acronym: PICTURE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-189-03
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Results first posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging (Experimental): General imaging subjects receiving CT exams
  Interventions: Device: 64 Channel VCT

INTERVENTIONS:
Device: 64 Channel VCT — cardiac CT angiography exam

SUMMARY:
To determine the relative efficacy of Cardiac Computed Tomography Angiography (CCTA) and Single Positron Emission Computed Tomography (SPECT) in patients with an intermediate risk of CAD.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, within-subject comparative study. One hundred fifty (150) subjects with CATH procedures are needed in the study. Approximately 300 subjects who meet all of the inclusion/exclusion criteria will be enrolled. The study population will consist of subjects with symptoms suspected of and at intermediate-risk for ischemic heart disease, which are referred for MPS for a definitive diagnosis of CAD.

Each subject will undergo the following procedures:

* A Myocardial Perfusion Study (MPS) procedure, as standard of care;
* An IV contrast-enhanced cardiac CT (CCTA) procedure;
* A CATH procedure when the MPS and/or cardiac CT examination is deemed positive or equivocal and at the discretion of the referring physicians, as a standard-of-care procedure.

When both the MPS and CCTA are normal, the subject is not required to undergo a CATH procedure, but will enter into follow-up. The research staff at each site will perform follow-up for each subject at 12 months (± 15 days) and 24 months (± 15 days) and 36 months (± 15 days) after the completion of the cardiac CT procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an intermediate probability risk for coronary artery disease.
* Subject has symptoms of suspected ischemic heart disease.
* Subject is at intermediate risk for coronary artery disease

Exclusion Criteria:

* The subject has undergone a prior CCTA within 6 months prior to entering the study.
* The subject has a documented history of CAD by CATH, myocardial infarction (MI), metal stent placement in any of the coronary vessels, or a previous coronary artery bypass graft (CABG) procedure
* The subject has hemodynamic or active clinical instability:

  * Acute chest pain (sudden onset);
  * Cardiac shock;
  * Unstable blood pressure (BP);
  * Severe congestive heart failure or acute pulmonary edema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Budoff, Study Chair — LA Biomedical Research Institute
Locations (1):
- GE Healthcare, Waukesha, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Imaging: Enrolled subjects for general imaging
Period: Overall Study
Arm/Group | Imaging
Started | 249
Completed | 249
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects
Arm/Group | Imaging
Number analyzed (Participants) | 249
Age, Continuous [Mean (Full Range); unit: years] | 30 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender was not record for analysis for this study.

OUTCOME MEASURES:

1. Primary Outcome: Detection of Significant Coronary Artery Disease Using Diagnostic Catheterization for Standard of Truth.
Description: Number of subjects with CT for detection purposes
Time Frame: through study completion, an expected average of 1 year
Population: Data were not collected for analysis.
Groups:
- Enrolled: Enrolled subjects for general imaging
Arm/Group | Enrolled
Number analyzed (Participants) | 0
Value | 0

2. Secondary Outcome: Clinical Outcomes - EKG, Laboratory Workup, Changes in Medical Management, Downstream Cardiac Testing, Significant Coronary Interventions, and Major Cardiac Events & Long-term Outcomes (Non-fatal MI and Cardiac-related Death).
Time Frame: 1 year outcomes after initial MPS exam
Population: Data were not collected for analysis.
Groups:
- Outcome Measure 2: 1 year clinical outcome follow-up (Study terminated prior to collection)
Arm/Group | Outcome Measure 2
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Groups:
- Enrolled: Subjects receiving diagnostic CT scans
Arm/Group | Enrolled
Serious Adverse Events (participants affected / at risk) | 0/249
Other Adverse Events (participants affected / at risk) | 0/249

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No